CLINICAL TRIAL: NCT03592667
Title: Effect of Dapagliflozin on the Blood Pressure Variability and the Ambulatory Arterial Stiffness Index in Individuals With Stage I Hypertension Without Diabetes Mellitus
Brief Title: Dapagliflozin on Blood Pressure Variability and Ambulatory Arterial Stiffness Index in Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Professor investigator titular C, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAPA on VBP-AASI Hypertension
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-08

CONDITIONS: Hypertension
Keywords: Stage I Hypertension; Without type 2 diabetes mellitus; Variability of blood pressure; Ambulatory arterial stiffness index; Dapagliflozin; ABPM
MeSH Terms: conditions — Hypertension | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin capsules, 10 mg, one per day before breakfast during 12 weeks.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo capsules, one per day before breakfast during 12 weeks.
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg, one per day before breakfast during 12 weeks.
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo - Cap — One per day before breakfast during 12 weeks.
  Other Names: Calcined magnesium
  Arms: Placebo

SUMMARY:
The prevalence of arterial hypertension has remained the same in the last 5 years, however, almost 50% of the population continues without an adequate adjustment according to the National Health Survey of the Midway 2016.

It has been shown that the variability of blood pressure (VBP) during 24 h and visit-visit is associated with cardiovascular diseases (CVD) over the effect of blood pressure (BP) itself. On the other hand, arterial stiffness is well known as an independent factor of CVD risk and for its evaluation the ambulatory arterial stiffness index (AASI) has been proposed. AASI and the VPA obtained through an evaluation by ambulatory BP monitoring (ABPM) individual of 24 h.

Dapagliflozin is an inhibitor of the sodium-glucose cotransporter type 2 (iSGLT2) for the treatment of diabetes mellitus type 2 (DM2) that promotes natriuresis and osmotic diuresis, which produces a decrease in plasma volume and a decrease in BP.

The aim of ths study is to evaluate the effect of dapagliflozin on VBP and AASI in individuals with stage I hypertension whitout DM2.

The investigators hypothesis is that the administration of dapagliflozin decreases the VBP and AASI in individuals with stage I hypertension whitout DM2.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial in 20 patients with a diagnosis of stage I hypertension without DM2.

They will be assigned randomly two groups of 10 patients each to receive 10 mg of Dapagliflozin (Forxiga, Astra Zeneca) or placebo, one per day before breakfast during 12 weeks.

There will be calculated indices of VBP: 24 h, daytime and night-time standard deviation (SD), coefficient of variation (CV), 24 h weighted SD, Day-to-nigth BP changes and average real variability (AVR). On the other hand, AASI will be calculated with a linear regression.

This protocol it's already approved by the local ethics committee and written informed consent it's going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentages for variable qualitative. Qualitative variables will be analyzed by X2 o exact fisher test, will be used for differences inter-group. Mann-Whitney U Test and Wilcoxon Test for the within-groups differences. It will be considered statistical significance p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patients both sexes, age between 30 and 60 years
* Diagnosis of stage I hypertension according ACC/AHA (American college of cardiology/American heart association) blood pressure between 130-139/ 80-89 mmHg.
* Fasting plasma glucose < 100 mg/dl
* BMI >35 kg/m2
* Glomerular filtration rate > 60ml/min/1.73m2

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to ingredients of intervention
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart, thyroid or cardiovascular diseased
* Previous treatment for hypertension or depression
* Triglycerides ≥ 400 mg/dl
* Total cholesterol ≥ 240 mg/dl
* Worker per shift night
* Arrhythmia

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Indices of blood pressure: 24 h, daytime and night-time SD and CV, 24 h weighted SD, day-to-nigth BP changes and ARV | Baseline to Week 12
  Blood pressure variability will be evaluated with ambulatory blood pressure monitoring
Ambulatory arterial stiffness index | Baseline to Week 12
  Arterial stiffness will be evaluated with ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Pulse Pressure of 24 h | Baseline to Week 12
  Will be evaluated with ambulatory blood pressure monitoring, systolic BP minus diastolic BP.
Mean arterial pressure of 24 h, daytime and nigth-time | Baseline to Week 12
  Will be evaluated with ambulatory blood pressure monitoring, systolic BP minus diastolic BP/3, plus diastolic BP.
Heart rate of 24 h, daytime and nigth-time | Baseline to Week 12
  Will be evaluated with ambulatory blood pressure monitoring.
Hypertensive load daytime and nigth-time | Baseline to Week 12
  Will be evaluated with ambulatory blood pressure monitoring.
White coat hypertension | Baseline to Week 12
  will be evaluated with ambulatory blood pressure monitoring
Fasting glucose levels | Baseline to Week 12
  The fasting glucose levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 12.
Total cholesterol | Baseline to Week 12
  Total cholesterol levels will be evaluated at baseline and week 12 by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at week 12
Triglycerides levels | Baseline to Week 12
  Triglycerides levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at week 12
High density lipoprotein (c-HDL) levels | Baseline to Week 12
  c-HDL levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at week 12
Creatinine levels | Baseline to Week 12
  Creatinine levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques
Uric acid levels | Baseline to Week 12
  Uric acid levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques
Body Weight | Baseline, week 4, week 8 and week 12
  The body weight will be measured at baseline, week 4, week 8 and week 12 with a bioimpedance balance and the entered values reflect the body weight at week 12
Body Mass Index | Baseline, week 4, week 8 and week 12
  Body Mas Index will be calculated at baseline, week 4, week 8 and week 12 with the Quetelet index formula and the entered values reflect the body mass index at week 12
Waist circumference | Baseline, week 4, week 8 and week 12
  Waist circumference will be evaluated with the method proposed by ISAK.
Glomerular filtration rate | Baseline to Week 12
  Glomerular filtration rate will be calculated at baseline and week 12 with the Cockcroft-Gault formula and the entered values reflect the Glomerular filtration rate at week 12

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico